CLINICAL TRIAL: NCT06853613
Title: Effects of an Adapted Multicomponent Training Program (Adapted Physical and Sports Activity - AFA) for Promoting Mental and Physical Well-being in Cancer Survivors Currently in Physiological or Chronic-stabilized Condition
Brief Title: Comparing Multicomponent and Aerobic Training: Impact on Fitness, Psychological and Quality of Life Parameters in Cancer Survivors Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Luca Poli, Dr., University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0324886
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cancer Survivors
Keywords: cancer-related fatigue; mental and physical well-being; muscle function; anxiety-depressive symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multicomponent Training (MCT) (Experimental): subjects assigned to the MCT group will perform a training protocol defined multicomponent training, which includes aerobic, resistance and flexibility components.
  Interventions: Other: Multicomponent Training Protocol
- Aerobic training (AT) (Experimental): subjects assigned to the AT group will perform training protocol of only aerobic exercises.
  Interventions: Other: Aerobic Training Protocol
- Waiting List Control Group (WLCG) (No Intervention): Subjects assigned to the WLCG group will not engage in any structured physical activity throughout the intervention period, continuing with their usual lifestyle, and will be placed on a waiting list, ensuring their participation in adapted physical activity at the end of the 24-week intervention.

INTERVENTIONS:
Other: Multicomponent Training Protocol — Each session consists of:
  Warm-up (10 minutes): Low-intensity walking (Borg scale 10-11) to increase heart rate, improve blood flow, and prepare joints.
  Main phase (40 minutes):
  Aerobic exercises: Controlled jumping jacks, step-ups, alternating knee lifts, lateral steps, and leg lifts.
  Mobility exercises: Thoracic extensions, cat-to-cows, overhead stretching with a stick, and hip internal rotations (1-3 sets, 30-60 seconds per exercise).
  Resistance training: Gradual progression of 8 exercises targeting major muscle groups, such as squats, bicep curls, shoulder presses, and rows (1-3 sets, 10-15 reps, RPE 13-15).
  Cool-down (10 minutes): Breathing exercises and stretching (1-3 sets, 10-30 seconds per stretch).
  Arms: Multicomponent Training (MCT)
Other: Aerobic Training Protocol — Each training session will include an initial 10-minute muscle activation phase (low-intensity walking, Borg = 10-11) to increase heart rate, improve muscle blood flow, and prepare the major joints for the next work phase.
  main exercise period (40-minute):
  25 minutes of progressive aerobic exercises (controlled and rhythmic jumping jacks, step-ups on a sturdy platform (such as a low step or stable surface), standing knee raises (alternating legs), fast side steps or side leg raises).
  15 minutes of walking, exercises will be performed at an intensity to ensure that perceived exertion (RPE) will remain between 13 and 15 points on the Borg Scale (6-20). Progression over the weeks will be by maintaining intensity in this range.
  Cool down period: breathing and stretching exercises on all major muscle groups.
  Arms: Aerobic training (AT)

SUMMARY:
The goal of this clinical trial is to evaluate if a multicomponent training program (MCT), including aerobic and resistance exercises, or an aerobic training program (AT) can improve physiological, physical fitness, mental well-being, and quality of life in cancer survivors currently stabilized. The main questions it aims to answer are:

Does MCT or AT improve physiological parameters, physical fitness, mental well-being, and overall quality of life compared to a waitlist control group (WLCG)? Does MCT provide superior physiological an psychological improvements compared to AT?

Researchers will compare:

MCT (a combination of aerobic, mobility, and resistance training exercises) AT (an aerobic-solo training) to see if these interventions improve fitness, health, psychological and quality of life outcomes compared to WLCG (participants not engaging in structured physical activity during the study), and if there will be significant differences between MCT and AT .

Participants will:

Complete assessments of anthropometric, physical fitness, and psychological parameters at baseline (T0) and after 24 weeks (T1).

Be randomly assigned to one of three groups (MCT, AT, or WLCG).

Engage in a 24-week structured training program (MCT or IMCT) supervised by exercise professionals, including:

Warm-up sessions (10 minutes, low-intensity walking). Main sessions (40 minutes): aerobic, mobility, resistance (MCT), only-aerobic (AT) exercises.

Cool-down sessions (10 minutes): breathing and stretching exercises.

This study will provide insights into the efficacy of tailored physical activity interventions for stabilized Cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Women/Men;
* Age between 18 and 80 years at the time of initial treatment;
* Subjects in remission for at least 3 months;
* No diagnosis of secondary cancer at baseline;
* No physical impediment to physical activity (Eastern Cooperative Oncology Groups (ECOG) performance status 0-1);
* Signature of a written informed consent form (or their legally recognized representatives must sign) indicating that the patient understood the purpose and procedures required for the study and is willing to participate in the study;
* Sedentary lifestyle (subjects who have not followed WHO guidelines for aerobic and resistance exercise in the past 3 months).
* Currently in treatment, as long as not hospitalized, in stabilized chronic condition,
* Positive medical specialist assessment of noncompetitive physical activity practice.

Exclusion Criteria:

* Metastasis;
* Uncontrolled hypertension or untreated heart disease;
* Severe musculoskeletal or joint disorders with severe mobility limitations;
* Psychiatric disorders;
* Taking psychotropic drugs;
* Inability to engage in physical activity;
* Lack of fitness to practice sports.
* Expected absence of more than two weeks during the intervention period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Body body fat percentage | 24-weeks
  Body fat percentage assessed throught the Bioelectrical Impedance Analysis (BIA):
  Body fat percentage (in %)
  The procedure involves sending a low-level electrical current through the body and measuring resistance.
  Interpretation:
  Higher body fat percentage indicates more fat.
Change in Body Water | 24-weeks
  Body water content assessed throught the Bioelectrical Impedance Analysis (BIA):
  Total body water (in %)
  The procedure involves sending a low-level electrical current through the body and measuring resistance.
  Interpretation:
  Higher total body water suggests better hydration.
Change in Muscle Mass | 24-weeks
  muscle mass assessed throught the Bioelectrical Impedance Analysis (BIA):
  Muscle mass (in kg)
  The procedure involves sending a low-level electrical current through the body and measuring resistance.
  Interpretation:
  Higher muscle mass suggests better muscle development.
Change in lower body strength | 24-weeks
  30-s chair stand (30CST) test: Sit-to-stand from a chair during 30 seconds (measured in seconds)
Change in functional mobility | 24-weeks
  Timed Up and Go (TUG) Test (measured in seconds)
Change in Handrigp Strength | 24-weeks
  Handgrip Strength (HGS) test: muscle strength measured with manual dynamometers (Kgf)
Change in aerobic capacity | 24-weeks
  2-Minute Step Test (TMST): march in place for 2 minutes, lifting their knees to a height halfway between the iliac crest and the patella.The number of full knee lifts (repetitions) completed in 2 minutes is recorded.
Change in lower body flexibility | 24-weeks
  Chair Sit-and-Reach Test: measures lower body flexibility (hamstrings and lower back) in centimeters (cm). It involves sitting on a chair, extending one leg, and reaching toward the toes to assess mobility. The measurement is taken by recording the distance between the fingertips and the toes. Positive score (+): Fingertips go past the toes.Zero score (0): Fingertips touch the toes. Negative score (-): Fingertips fall short of the toes.
  A ruler or tape measure is used to record the exact distance.
Change in upper body flexibility | 24-weeks
  Back Scratch Test: measures upper body flexibility, particularly shoulder mobility, in centimeters (cm). It involves reaching one hand over the shoulder and the other behind the back to touch or overlap fingers.
  Positive score (+): Fingers overlap (measured as the overlap distance). Zero score (0): Fingers just touch. Negative score (-): Fingers do not touch (measured as the gap distance).
  A ruler or tape measure is used to record the exact distance.
Change in psychological parameters (anxiety). | 24-weeks
  State-Trait Anxiety Inventory (STAI-Y): measures anxiety levels using a numerical score. It consists of 20 items assessing temporary (state) anxiety on a 4-point scale (1 = not at all to 4 = very much so).
  Total score range: 20 to 80 (higher scores indicate greater anxiety).
  Interpretation:
  20-37: Low anxiety 38-44: Moderate anxiety 45-80: High anxiety
  The final score is obtained by summing the responses.
Change in psychological parameters (depression). | 24-weeks
  Beck Depression Inventory (BDI): measures depression severity using a numerical score. It consists of 21 items, each rated on a 4-point scale (0 to 3) based on symptom severity.
  Total score range: 0 to 63 (higher scores indicate more severe depression).
  Interpretation:
  0-13: Minimal depression 14-19: Mild depression 20-28: Moderate depression 29-63: Severe depression
  The final score is obtained by summing the responses.
Change in psychological parameters (Fatigue). | 24-weeks
  Fatigue Severity Scale (FSS): measures the impact of fatigue on daily life using a numerical score. It consists of 9 items, each rated on a 7-point scale (1 = strongly disagree to 7 = strongly agree).
  Total score range: 9 to 63 (higher scores indicate greater fatigue severity).
  Interpretation:
  * 36: Low to moderate fatigue >36: High fatigue
  The final score is the average of all 9 responses.
Change in psychological parameters (Quality of Life). | 24-weeks
  EORTC QLQ-C30: assesses the quality of life in cancer patients using a numerical score. It consists of 30 questions covering functional status, symptoms, and overall health, rated on a 4-point scale (1 = not at all to 4 = very much) or a 7-point scale (1 = very poor to 7 = excellent).
  Scores range from 0 to 100 (higher scores indicate better functioning for global health/function scales and worse symptoms for symptom scales).
  Interpretation:
  Functional scales: Higher scores = better function. Symptom scales: Higher scores = more severe symptoms.
  Scores are calculated and standardized based on EORTC guidelines.
Change in psychological parameters (Coping). | 24-weeks
  Brief COPE: assesses coping strategies using a numerical score. It consists of 28 items, grouped into 14 coping strategies, each rated on a 4-point scale (1 = I haven't been doing this at all to 4 = I've been doing this a lot).
  Scores range from 2 to 8 per coping strategy (higher scores indicate greater use of that coping strategy).
  Interpretation:
  Higher scores in adaptive strategies (e.g., active coping, planning) suggest positive coping.
  Higher scores in maladaptive strategies (e.g., denial, self-blame) may indicate ineffective coping.
  Final scores are analyzed per strategy rather than as a total score.

SECONDARY OUTCOMES:
Evaluation of adherence to training protocols | 24-weeks
  Adherence (%): (Number of prescribed activities/Number of completed activities )×100

CONTACTS AND LOCATIONS:
Overall Officials: Luca Poli, Dr., Principal Investigator — University of Bari Aldo Moro
Locations (1):
- Società Ginnastica Angiulli, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT06853613/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT06853613/ICF_001.pdf